CLINICAL TRIAL: NCT02599922
Title: A Multiple-Site, Phase 1/2, Safety and Efficacy Trial of a Recombinant Adeno-associated Virus Vector Expressing CNGB3 in Patients With Congenital Achromatopsia Caused by Mutations in the CNGB3 Gene
Brief Title: Safety and Efficacy Trial of AAV Gene Therapy in Patients With CNGB3 Achromatopsia (A Clarity Clinical Trial)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGTC_CNGB3-001; R24EY022023 (NIH)
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Achromatopsia
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Group 1: 2.0 x 10^11 vg/mL of AGTC-401 (Experimental): Subjects at least 18 y/o treated with 2.0 x 10^11 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 2: 4.0 x 10^10 vg/mL of AGTC-401 (Experimental): Subjects at least 18 y/o treated with 4.0 x 10^10 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 3: 1.2 x 10^11 vg/mL of AGTC-401 (Experimental): Subjects at least 18 y/o treated with 1.2 x 10^11 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 4: 3.6 x 10^11 vg/mL of AGTC-401 (Experimental): Subjects at least 18 y/o treated with 3.6 x 10^11 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 4a: 3.6 x 10^11 vg/mL of AGTC-401 (Experimental): Subjects 6 to 17 y/o treated with 3.6 x 10^11 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 5: 1.1 x 10^12 vg/mL of AGTC-401 (Experimental): Subjects at least 18 y/o treated with 1.1 x 10^12 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 5a: 1.1 x 10^12 vg/mL of AGTC-401 (Experimental): Subjects 4 to 8 y/o treated with 1.1 x 10^12 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 6: 3.2 x 10^12 vg/mL of AGTC-401 (Experimental): Subjects at least 18 y/o treated with 3.2 x 10^12 vg/mL of rAAV2tYF-PR1/7-hCNGB3 study drug.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3
- Group 7: MTD of AGTC-401 (Experimental): Subjects 4 to 8 y/o treated with a maximum tolerated dose of rAAV2tYF-PR1/7-hCNGB3 study drug determined by Groups 1-6.
  Interventions: Biological: rAAV2tYF-PR1.7-hCNGB3

INTERVENTIONS:
Biological: rAAV2tYF-PR1.7-hCNGB3 — rAAV2tYF-PR1.7-hCNGB3 is a non-replicating, rep/cap-deleted, recombinant adeno-associated virus vector that expresses the CNGB3 gene.
  Other Names: AGTC-401

SUMMARY:
This will be a non-randomized, open-label, Phase 1/2 study of the safety and efficacy of AGTC-401 administered to one eye by subretinal injection in individuals with achromatopsia caused by mutations in the CNGB3 gene. The primary study endpoint will be safety and the secondary study endpoint will be efficacy.

DETAILED DESCRIPTION:
This will be a non-randomized, open-label, Phase 1/2 study of the safety and efficacy of AGTC-401 administered to one eye by subretinal injection in individuals with achromatopsia caused by mutations in the CNGB3 gene. The primary study endpoint will be safety and the secondary study endpoint will be efficacy.

Subjects will be enrolled sequentially in seven dosing groups. Subjects in Groups 1, 2, 3, 4, 5, and 6 will be at least 18 years of age and will receive varying dose levels of study agent. Subjects in Group 4a will be 6 to 17 years of age and will receive the same dose as Group 4. Subjects in Groups 5a and 7 will be between 4 and 8 years of age. Subjects in Group 5a will receive the same dose as Group 5, and subjects in Group 7 will receive the maximum tolerated dose identified in Groups 1, 2, 3, 4, 4a, 5, 5a, and 6.

Safety will be monitored by evaluation of ocular and non-ocular adverse events and hematology and clinical chemistry parameters. Efficacy parameters will include visual acuity, light discomfort testing, color vision, static visual field, ERG, adaptive optics retinal imaging, functional MRI (fMRI), color brightness test and OCT.

ELIGIBILITY:
Inclusion Criteria include:

1. Male or female subjects with documented mutations in both alleles of the CNGB3 gene;
2. Retinal disease consistent with a clinical diagnosis of achromatopsia;
3. At least 18 years of age for Groups 1, 2, 3, 4, 5 and 6. At least 6 years of age for Group 4a, and 4-8 years of age for Groups 5a and 7;
4. Able to perform tests of visual and retinal function;
5. Visual acuity in the study eye not better than 55 ETDRS letters (Snellen equivalent 20/80) based on the average of two examinations at the baseline visit;
6. Acceptable laboratory parameters;
7. For females of childbearing potential: A negative pregnancy test within 2 days before administration of study agent.

Exclusion Criteria include:

1. Best-corrected visual acuity difference between the two eyes of > 15 ETDRS letters (3 lines);
2. Evidence of degenerative myopia in the study eye;
3. Pre-existing eye conditions that would contribute to vision loss in either eye or increase the risk of subretinal injection in the study eye.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 year
  Proportion of participants experiencing grade 3 or greater adverse events

SECONDARY OUTCOMES:
Visual acuity | 1 year
  Changes in best corrected visual acuity compared to pre-treatment
Light aversion | 1 year
  Changes in light discomfort testing compared to pre-treatment
Color vision | 1 year
  Changes in color vision testing compared to pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Jacobs, MD, MBA, Study Director — Applied Genetic Technologies Corporation
Locations (8):
- United States (8):
  - VitreoRetinal Associates, Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Pangere Center for Inherited Retinal Diseases, The Chicago Lighthouse for People Who Are Blind or Visually Imp, Chicago, Illinois
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke Eye Center, Duke University Medical Center, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Casey Eye Institute, Oregon Health and Sciences University, Portland, Oregon

REFERENCES:
- [Background] Komaromy AM, Alexander JJ, Rowlan JS, Garcia MM, Chiodo VA, Kaya A, Tanaka JC, Acland GM, Hauswirth WW, Aguirre GD. Gene therapy rescues cone function in congenital achromatopsia. Hum Mol Genet. 2010 Jul 1;19(13):2581-93. doi: 10.1093/hmg/ddq136. Epub 2010 Apr 8. PMID 20378608
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931
- See also: Sponsor website — http://www.agtc.com